CLINICAL TRIAL: NCT06114368
Title: Outcomes Evaluation of Endoscopic Flexor Hallucis Longus Transfer Versus Minimally Invasive Primary Repair in Patients With Acute Achilles Tendon Rupture
Brief Title: Endoscopic Flexor Hallucis Longus Transfer vs Minimally Invasive Repair in Acute Achilles Tendon Rupture
Status: Enrolling by invitation | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: General Hospital of Naoussa (Unknown); Private Orthopedics Practice P. Symeonidis (Unknown)
Responsible Party: Principal Investigator, Michail Kotsapas, Michail Kotsapas, MD, MSc, Resident of Orthopedics (General Hospital of Naoussa), PhD Candidate (Aristotle University of Thessaloniki), Aristotle University Of Thessaloniki
Other Study IDs: 26543
Record Dates: First submitted 2023-10-28; First posted 2023-11-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Achilles Tendon Rupture; Achilles Tendon Surgery; Achilles Tendon Injury
Keywords: Achilles tendon; rupture; Endoscopic; Flexor Hallucis Longus transfer; repair; Percutaneous Achilles Repair System - PARS; Minimally invasive
MeSH Terms: conditions — Rupture | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endoscopic Flexor Hallucis Longus transfer / Group 1: Patients with acute Achilles tendon rupture managed with Endoscopic Flexor Hallucis Longus transfer by one surgeon (A.E.) in one hospital (General Hospital of Naoussa, Naoussa, Greece), all of which followed the same rehabilitation protocol.
  Interventions: Procedure: Surgery for the treatment of Acute Achilles tendon rupture
- Minimally Invasive Primary repair / Group 2: Patients with acute Achilles tendon rupture managed with Minimally Invasive Primary repair by one surgeon (P.S.) in one hospital (St. Luke's Hospital, Thessaloniki, Greece), all of which followed the same rehabilitation protocol.
  Interventions: Procedure: Surgery for the treatment of Acute Achilles tendon rupture

INTERVENTIONS:
Procedure: Surgery for the treatment of Acute Achilles tendon rupture — Two different surgical techniques were applied in two different patient groups for the same disease. Their outcomes are evaluated and compared

SUMMARY:
The goal of this observational study is to compare the outcomes of two different surgical techniques (Endoscopic Flexor Hallucis Longus transfer - Group 1 vs Minimally Invasive primary repair - Group 2) for patients with acute Achilles tendon rupture. The main questions to be answered are:

1. Which group's patients are more satisfied?
2. Which group's patients appear to have a greater complication rate?
3. Which group's patients have greater calf and ankle circumference compared to the unaffected limb?
4. Which group's patients have greater passive and active range of ankle motion compared to the unaffected limb?
5. Are group 1 patients characterized by strength deficit in hallux flexion power?

DETAILED DESCRIPTION:
Two separate foot and ankle surgeons in Northern Greece prefer to use a different surgical technique in their respective patients with Acute Achilles tendon rupture.

The first one (A.E.) prefers to perform only Endoscopic Flexor Hallucis Longus transfer, while the second one (P.S.) prefers to perform only Minimally invasive primary repair assisted by the Achillon device (Percutaneous Achilles Repair System - PARS). They both agreed to enroll their recently operated patients (last 5 years) in this retrospective study, which will be conducted by the researcher (M.K.). The patient's study may be retrospective, nevertheless, the patients were randomly chosen and enrolled by a prospectively designed study protocol. Each surgeon applied the respective surgical treatment modality regardless of each patient's characteristics, biometrics, or comorbidities. Inclusion and Elimination criteria will be applied. The patient's satisfaction will be evaluated with the Achilles Tendon Total Rupture Score (ATRS). Complications will be documented. Calf and ankle circumference will be measured and compared to the contralateral healthy limb. Ankle passive and active range of motion will be measured and compared to the contralateral healthy limb. Possible correlations will be investigated regarding patient age, BMI, history of smoking, level of activity, and comorbidities.

ELIGIBILITY:
Inclusion Criteria:

* Signed Consent Form
* Age between 18-75 years
* Acute Achilles Tendon Rupture (<3 weeks)
* Surgical Management with Endoscopic Flexor Hallucis Longus transfer or Minimally Invasive primary tendon repair
* More than 12 months postoperative follow-up
* Patients operated after 2015

Exclusion Criteria:

* Inability or Unwillingness to cooperate
* Medically unfit for examination (e.g. due to terminal illness)
* Age less than 18 or more than 75 years
* Non-operative Management as definitive treatment
* Surgical Management other than the ones described in the inclusion criteria
* Neglected Achilles Tendon Rupture (>3 weeks)
* Bilateral Achilles Tendon Rupture
* Patients operated before 2015
* Comorbidities interfering with the secondary outcomes (e.g. Venous insufficiency resulting in lower limb excessive edema interferes with ankle and calf circumference, rheumatoid arthritis and/or previous foot and ankle surgery interferes with active and passive range of motion of the ankle, etc)

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with Achilles tendon rupture operated exclusively with these two surgical techniques, by these two particular surgeons (A.E. and P.S.) in their respective hospitals (General Hospital of Naoussa, St Luke's Hospital).
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-03-05 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction assessed with the Achilles Tendon Total Rupture Score | More than 12 months postoperatively
  Evaluated and quantified with the Achilles Tendon Total Rupture Score (minimum value = 0 - worst outcome, maximal value = 100 - best outcome)

SECONDARY OUTCOMES:
Complication Rate | More than 12 months postoperatively
  Complications will be recorded and categorized: Rerupture, Infection, Nerve injury, Miscellaneous
Calf Circumference | More than 12 months postoperatively
  Calf circumference measured 15 cm distally to the inferior pole of the patella. Contralateral limb calf circumference will also be measured. The Calf Circumference Difference will be calculated and compared between the two groups.
Ankle Circumference | More than 12 months postoperatively
  Ankle circumference measured 8 cm proximally to the lateral malleolus. Contralateral limb ankle circumference will also be measured. The Ankle Circumference Difference will be calculated and compared between the two groups.
Ankle joint Range of Motion | More than 12 months postoperatively
  Active and Passive Ankle joint Range of Motion will be calculated with an electronic goniometer. Contralateral limb Range of Ankle joint Motion will also be measured. The Range of Motion Difference will be calculated and compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Michail K. Kotsapas, MD, MSc, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- General Hospital of Naoussa, Náousa, Central Macedonia, Greece

IPD SHARING:
Plan to Share IPD: Undecided
The records of each patient to be enrolled belong to the respective surgeon (A.E. and P.S.). Thus, the records of each patient will be entrusted to the main researcher (M.K.) with the obligation to maintain doctor-patient confidentiality. The final study results will not reveal any sensitive patient data (de-identification). Photos and videos of each patient's examination may be taken after ensuring their written and oral informed consent.

REFERENCES:
- [Result] Abdelatif NMN, Batista JP. Outcomes of Percutaneous Achilles Repair Compared With Endoscopic Flexor Hallucis Longus Tendon Transfer to Treat Achilles Tendon Ruptures. Foot Ankle Int. 2022 Sep;43(9):1174-1184. doi: 10.1177/10711007221096674. Epub 2022 Jun 10. PMID 35686445
- [Result] Abdelatif NMN, Batista JP. Endoscopic Flexor Hallucis Longus Transfer for the Management of Acute Achilles Tendon Ruptures in Professional Soccer Players. Foot Ankle Int. 2022 Feb;43(2):164-175. doi: 10.1177/10711007211036439. Epub 2021 Sep 24. PMID 34558318
- [Result] Batista JP, Abdelatif NMN, Del Vecchio JJ, Diniz P, Pereira H. Endoscopic Flexor Hallucis Longus Transfer for the Management of Acute Achilles Tendon Ruptures: A Prospective Case Series Report With a Minimum of 18 Months' Follow-Up. J Foot Ankle Surg. 2020 Sep-Oct;59(5):927-937. doi: 10.1053/j.jfas.2019.12.008. Epub 2020 Jun 9. PMID 32527698
- [Result] Martin KD, Crouser NJ, Khan IA. Minimally Invasive Mid-Substance Achilles Tendon Repair Using the Percutaneous Achilles Repair System (PARS). JBJS Essent Surg Tech. 2022 Sep 22;12(3):e21.00050. doi: 10.2106/JBJS.ST.21.00050. eCollection 2022 Jul-Sep. PMID 36816527